CLINICAL TRIAL: NCT01472159
Title: Optimizing CGM Use and Metabolic Outcomes in Youth With Type 1 Diabetes
Brief Title: Can Glucose Monitoring Improve (CGMi Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Jaeb Center for Health Research (Other)
Responsible Party: Principal Investigator, Lori Laffel, Chief, Pediatric, Adolescent, & Young Adult Section; Investigator, Genetics & Epidemiology Section, Joslin Diabetes Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-28; R01DK089349 (NIH)
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CGM-Usual Care (No Intervention): * Routine CGM education
- CGM-Teamwork (Experimental): * Routine CGM education
  * CGM Family Teamwork Intervention
  Interventions: Behavioral: CGM Family Teamwork Intervention

INTERVENTIONS:
Behavioral: CGM Family Teamwork Intervention — The family-focused behavioral intervention targets barriers associated with sustained CGM use in youth with type 1 diabetes. During months 1-18, families in the intervention group will participate in the intervention at each study visit for about an additional 30 minutes.
  Arms: CGM-Teamwork

SUMMARY:
The purpose of this 2-year randomized controlled trial (RCT) is to implement and evaluate a family-focused behavioral teamwork intervention aimed at overcoming barriers to sustained continuous glucose monitoring (CGM) use in youth with type 1 diabetes (T1D). We hypothesize that CGM implemented with a family-focused, behavioral teamwork intervention will result in sustained CGM use and greater improvement in A1c compared to routine implementation of CGM.

DETAILED DESCRIPTION:
Consistent CGM use in youth with T1D has been difficult to sustain historically. Youth with T1D and their families have routinely felt burden related to the introduction of this technology into their care management. Additionally, there can be difficulties with calibration, skin irritation, frequent skips, excessive or nuisance alarms and inaccurate readings which often lead to diminished use or discontinuation entirely. The purpose of this protocol is to implement and evaluate a family-focused behavioral teamwork intervention aimed at overcoming barriers to sustained CGM use in youth with T1D. In this 2-year RCT, we will assess the long-term acceptability and durability of CGM use and its associated glycemic and psychological outcomes in youth with T1D and their families. We will randomize 120 families to one of two groups: (1) CGM implemented according to usual care (CGM-Usual Care, CGM-UC) or (2) CGM implemented with a family teamwork intervention (CGM-Teamwork, CGM-TW). This intervention will allow participants and families to overcome barriers to sustained CGM use and achieve glycemic benefits that have been afforded to adults using CGM as demonstrated in other research. In year 1, all CGM supplies will be provided and covered by study resources. In year 2, study participants will be asked to cover the costs associated with sensor use and any costs associated with replacement of CGM components in a manner consistent with routine clinical care as the investigators believe that it is important to assess durability of CGM use in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-17 years
* Planning to be living at home for 2 years
* Type 1 diabetes of at least 1 year duration
* Daily insulin dose ≥0.5 units/kg
* A1c ≥6.5% and ≤10.0%
* Insulin therapy with continuous subcutaneous insulin infusion (CSII) or multiple daily injections (≥3 injections/day)
* Blood glucose (BG) monitoring frequency ≥4 times/day
* Agreement to wear a CGM device
* Fluency in English for child and parent/guardian
* Stable living situation for ≥6 months (e.g., no Department of Youth Services Involvement)
* Joslin Clinic attendance: At least one Joslin Clinic visit in last year AND Anticipated care at Joslin Clinic for duration of study

Exclusion Criteria:

* Consistent CGM use, defined as 6+ days/week during the previous 6 months
* History of severe, life-threatening skin reactions to the adhesive used with the CGM device
* Pregnancy in the youth participant or intention to become pregnant within the next 2 years
* Significant developmental or cognitive disorder in the youth or parent/guardian that would prevent full participation in a family-based, behavioral intervention or implementation of CGM
* Inpatient psychiatric admission within the previous 6 months
* Participation in another intervention study during the previous 3 months
* Intent to enroll in another intervention study during the study period

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in glycemic control, assessed by hemoglobin A1c | Baseline and 1 year

SECONDARY OUTCOMES:
Change in psychosocial factors (e.g., self-efficacy, fear of hypoglycemia, quality of life, diabetes-specific family conflict, diabetes responsibility sharing, diabetes-specific burden, anxiety, depressive symptoms) | Baseline and 1 year
Change in glycemic control, assessed by hemoglobin A1c | 1 year and 2 years
  Durability of the intervention will be assessed by change in A1c from 1 year to 2 years
Change in psychosocial factors (e.g., self-efficacy, fear of hypoglycemia, quality of life, diabetes-specific family conflict, diabetes responsibility sharing, diabetes-specific burden, anxiety, depressive symptoms) | 1 year and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lori Laffel, MD, MPH, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] McGill DE, Volkening LK, Butler DA, Harrington KR, Katz ML, Laffel LM. Baseline Psychosocial Characteristics Predict Frequency of Continuous Glucose Monitoring in Youth with Type 1 Diabetes. Diabetes Technol Ther. 2018 Jun;20(6):434-439. doi: 10.1089/dia.2018.0037. Epub 2018 May 4. PMID 29727245
- [Result] Telo GH, Volkening LK, Butler DA, Laffel LM. Salient characteristics of youth with type 1 diabetes initiating continuous glucose monitoring. Diabetes Technol Ther. 2015 Jun;17(6):373-8. doi: 10.1089/dia.2014.0290. Epub 2015 Mar 6. PMID 25749206
- [Result] Volkening LK, Gaffney KC, Katz ML, Laffel LM. Recruitment Into a Pediatric Continuous Glucose Monitoring RCT. J Diabetes Sci Technol. 2017 Jan;11(1):100-107. doi: 10.1177/1932296816656208. Epub 2016 Jul 9. PMID 27340247
- [Result] Giani E, Snelgrove R, Volkening LK, Laffel LM. Continuous Glucose Monitoring (CGM) Adherence in Youth With Type 1 Diabetes: Associations With Biomedical and Psychosocial Variables. J Diabetes Sci Technol. 2017 May;11(3):476-483. doi: 10.1177/1932296816676280. Epub 2016 Nov 1. PMID 27807014